CLINICAL TRIAL: NCT01742286
Title: A Phase I, Open-label, Dose Escalation Study of LDK378 in Pediatric Patients With Malignancies That Have a Genetic Alteration in Anaplastic Lymphoma Kinase (ALK)
Brief Title: Phase I Study of LDK378 in Pediatric, Malignancies With a Genetic Alteration in Anaplastic Lymphoma Kinase (ALK)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLDK378X2103; 2012-002074-31 (EudraCT Number)
Record Dates: First submitted 2012-11-30; First posted 2012-12-05 (Estimated); Results first posted 2020-06-09 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-05

CONDITIONS: ALK-activated Tumors
Keywords: LDK378; Ceritinib; pediatric; malignancies; anaplastic lymphoma kinase; ALK; ALK-activated tumors; neuroblastoma; rhabdomyosarcoma; anaplastic large-cell lymphoma; inflammatory myofibroblastic tumor
MeSH Terms: conditions — Neoplasms; Neuroblastoma; Rhabdomyosarcoma; Lymphoma, Large-Cell, Anaplastic; Granuloma, Plasma Cell | interventions — ceritinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- LDK378 (Experimental): All participants were administered a single-agent LDK378 (Ceritinib) orally, once daily, continuously in fasted or fed conditions.
  Interventions: Drug: Ceritinib

INTERVENTIONS:
Drug: Ceritinib — LDK378 is a capsule taken by mouth, contents can be mixed with food for pediatric patients or mixed with water and given via nasogastric/gastric (NG/G) tube. For patients in fasted group: 1-2 tablespoons (15-30 mL) of an appropriate food such as apple sauce or non-fat yogurt and a glass of water were allowed.
  For patients in the fed cohort: LDK378 was taken with, or within 30 minutes after finishing a low-fat light snack containing 100-300 calories and 1.5-2 grams of fat.
  Other Names: LDK378

SUMMARY:
The purpose of this study was to estimate the maximum tolerated dose and/or recommended dose for expansion of LDK378 as a single agent, assess safety, tolerability and anti-tumor activity and characterize single and multiple-dose pharmacokinetics when administered orally to pediatric patients with ALK-activated tumors, with and without food.

DETAILED DESCRIPTION:
LDK378 is a novel inhibitor of ALK that is active in a broad range of ALK-activated tumor models, including models driven by mutated versions of ALK known to be resistant to crizotinib, and by ALK gene amplification.

The primary purpose of this study was to determine the maximum tolerated dose and/or recommended dose for expansion in pediatric patients, and to delineate a clinical dose to be used in any future pediatric studies, with and without food. This study also assessed the safety, tolerability, PK and preliminary evidence of antitumor activity of LDK378 in pediatric patients with neuroblastoma, and other ALK-activated tumors.

Fasted cohort: each daily dose of LDK378 (including days which involved PK blood sampling) was taken at least 2 hours after last meal & subjects did not eat until 1 hour after LDK378 was taken. Each daily dose of LDK378 was taken with 1-2 tablespoons (15-30 mL) of an appropriate food (such as applesauce or non-fat yogurt) & a glass of water

Fed cohort: each daily dose of LDK378 (including days which involved PK blood sampling) was taken with, or within 30 minutes after finishing a low-fat light snack containing 100-300 calories & 1.5-2 grams of fat.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with a locally advanced or metastatic malignancy that has progressed despite standard therapy, or for which no effective standard therapy exists
* Age ≥ 12 months and < 18 years
* The tumor must carry a genetic alteration of ALK
* Patients must have evaluable or measurable disease.
* Karnofsky performance status score ≥ 60% for patients > 12 years of age; Lansky score ≥ 50% for patients ≤ 12 years of age.

Exclusion criteria:

* Symptomatic central nervous system (CNS) metastases who are neurologically unstable or require increasing doses of steroids or local CNS-directed therapy (such as radiotherapy, surgery or intrathecal chemotherapy) to control their CNS disease
* Inadequate end organ function as defined by specified laboratory values
* Body surface area (BSA) < 0.35 m2
* Impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of LDK378 (e.g., ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, or malabsorption syndrome)
* Use of medications that are known to be strong inhibitors or inducers of CYP3A4/5 that cannot be discontinued at least 1 week prior to start of treatment with LDK378 and for the duration of the study
* Use of medications that are mainly metabolized by CYP3A4/5 or CYP2C9 that cannot be discontinued at least 1 week prior to start of treatment with LDK378 and for the duration of the study
* History of interstitial lung disease or interstitial pneumonitis, including clinically significant radiation pneumonitis
* History of pancreatitis or history of increased amylase or lipase that was due to pancreatic disease.
* Medications with a known risk of prolongation of QT interval

Ages: 12 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 83 (Actual)
Dates: Start 2013-08-28 (Actual); Primary Completion 2019-04-26 (Actual); Study Completion 2019-04-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (23):
- United States (5):
  - Dana Farber Cancer Institute Dept of Onc, Boston, Massachusetts
  - Memorial Sloan Kettering SC - 7, New York, New York
  - Cincinnati Children s Hospital Medical Center Dept of Oncology, Cincinnati, Ohio
  - St Jude s Childrens Research Hospital Dept of Oncology, Memphis, Tennessee
  - Texas Children's Hospital Dept of Oncology, Houston, Texas
- Australia (2):
  - Novartis Investigative Site, Randwick, New South Wales
  - Novartis Investigative Site, Parkville, Victoria
- Novartis Investigative Site, Toronto, Ontario, Canada
- France (2):
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Villejuif
- Germany (3):
  - Novartis Investigative Site, Cologne, North Rhine-Westphalia
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Essen
- Novartis Investigative Site, Milan, MI, Italy
- Netherlands (3):
  - Novartis Investigative Site, Utrecht, CS
  - Novartis Investigative Site, Amsterdam
  - Novartis Investigative Site, Rotterdam
- Novartis Investigative Site, Seoul, South Korea
- Spain (3):
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Valencia, Valencia
  - Novartis Investigative Site, Madrid
- United Kingdom (2):
  - Novartis Investigative Site, West Midlands, Birmingham
  - Novartis Investigative Site, Sutton, Surrey

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fischer M, Moreno L, Ziegler DS, Marshall LV, Zwaan CM, Irwin MS, Casanova M, Sabado C, Wulff B, Stegert M, Wang L, Hurtado FK, Branle F, Geoerger B, Schulte JH. Ceritinib in paediatric patients with anaplastic lymphoma kinase-positive malignancies: an open-label, multicentre, phase 1, dose-escalation and dose-expansion study. Lancet Oncol. 2021 Dec;22(12):1764-1776. doi: 10.1016/S1470-2045(21)00536-2. Epub 2021 Nov 12. PMID 34780709
- [Derived] Brivio E, Zwaan CM. ALK inhibition in two emblematic cases of pediatric inflammatory myofibroblastic tumor: Efficacy and side effects. Pediatr Blood Cancer. 2019 May;66(5):e27645. doi: 10.1002/pbc.27645. Epub 2019 Jan 29. PMID 30697903

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eighty-three patients were treated at different dose levels in both fasted and fed states dose escalation and expansion groups.
Pre-assignment Details: At least 15 patients for the fasted dose escalation & 12 patients for the fed dose escalation were expected to be treated. During the expansion part, approximately 45 patients were planned to be treated on the preferred regimen, approximately 25 patients in group 1 on the preferred regimen, and approximately 20 patients in group 2.
Groups:
- Fasted: Ceritinib 300 mg/m2: Participants in the fasted group who took 300 mg of ceritinib
- Fasted: Ceritinib 450 mg/m2: Participants in the fasted group who took 450 mg of ceritinib
- Fasted: Ceritinib 510 mg/m2: Participants in the fasted group who took 510 mg of ceritinib
- Fasted: Ceritinib 560 mg/m2: Participants in the fasted group who took 560 mg of ceritinib
- Fed: Ceritinib 320 mg/m2: Participants in the fed group who took 320 mg of ceritinib
- Fed: Ceritinib 400 mg/m2: Participants in the fed group who took 400 mg of ceritinib
- Fed: Ceritinib 500 mg/m2: Participants in the fed group who took 500 mg of ceritinib
Period: Escalation Phase
Arm/Group | Fasted: Ceritinib 300 mg/m2 | Fasted: Ceritinib 450 mg/m2 | Fasted: Ceritinib 510 mg/m2 | Fasted: Ceritinib 560 mg/m2 | Fed: Ceritinib 320 mg/m2 | Fed: Ceritinib 400 mg/m2 | Fed: Ceritinib 500 mg/m2
Started | 5 | 12 | 6 | 2 | 4 | 5 | 6
Ended Treatment = Not Completed) | 5 | 12 | 6 | 2 | 4 | 5 | 6
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 5 | 12 | 6 | 2 | 4 | 5 | 6
Not completed — Administrative problems | 1 | 1 | 0 | 0 | 0 | 0 | 2
Not completed — Adverse Event | 0 | 1 | 2 | 0 | 0 | 1 | 0
Not completed — Disease progression | 3 | 7 | 4 | 1 | 4 | 3 | 2
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Physician Decision | 0 | 3 | 0 | 1 | 0 | 0 | 2
Not completed — Subject/guardian decision | 1 | 0 | 0 | 0 | 0 | 0 | 0
Period: Expansion Phase
Arm/Group | Fasted: Ceritinib 300 mg/m2 | Fasted: Ceritinib 450 mg/m2 | Fasted: Ceritinib 510 mg/m2 | Fasted: Ceritinib 560 mg/m2 | Fed: Ceritinib 320 mg/m2 | Fed: Ceritinib 400 mg/m2 | Fed: Ceritinib 500 mg/m2
Started | 0 | 0 | 7 | 0 | 0 | 0 | 36
End of Treatment = Not Ccompleted | 0 | 0 | 7 | 0 | 0 | 0 | 36
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 7 | 0 | 0 | 0 | 36
Not completed — Administrative problems | 0 | 0 | 0 | 0 | 0 | 0 | 5
Not completed — Physician Decision | 0 | 0 | 4 | 0 | 0 | 0 | 9
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 6
Not completed — Disease progression | 0 | 0 | 3 | 0 | 0 | 0 | 15
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The Full analysis set (FAS) included all patients who received at least one dose of ceritinib.
Groups:
- Total: Total of all reporting groups
Arm/Group | Fasted: Ceritinib 300 mg/m2 | Fasted: Ceritinib 450 mg/m2 | Fasted: Ceritinib 510 mg/m2 | Fasted: Ceritinib 560 mg/m2 | Fed: Ceritinib 320 mg/m2 | Fed: Ceritinib 400 mg/m2 | Fed: Ceritinib 500 mg/m2 | Total
Number analyzed (Participants) | 5 | 12 | 13 | 2 | 4 | 5 | 42 | 83
Age, Continuous [Mean (Standard Deviation); unit: years] | 11.6 (5.27) | 10.0 (4.94) | 9.2 (5.34) | 9.0 (9.90) | 8.8 (4.99) | 9.2 (4.02) | 7.3 (4.73) | 8.5 (4.97)
Age, Customized [Number; unit: Participants]
  1 - < 7 yrs | 1 | 4 | 6 | 1 | 2 | 2 | 21 | 37
  7 - < 12 yrs | 2 | 2 | 1 | 0 | 0 | 1 | 10 | 16
  12 - < 18 yrs | 2 | 6 | 6 | 1 | 2 | 2 | 11 | 30
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 5 | 1 | 1 | 3 | 14 | 30
  Male | 2 | 9 | 8 | 1 | 3 | 2 | 28 | 53
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian | 0 | 1 | 1 | 0 | 0 | 0 | 3 | 5
  Black | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Caucasian | 5 | 7 | 11 | 2 | 4 | 3 | 33 | 65
  Other | 0 | 3 | 1 | 0 | 0 | 2 | 5 | 11
  Native American | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Incidence Rate of Dose Limiting Toxicities (DLTs) Occurring During First Cycle of Treatment
Description: A DLT is defined as an adverse event or abnormal laboratory value assessed as unrelated to disease, disease progression, inter-current illness, or concomitant therapies that occurs within the first 21 days of treatment with LDK378 and meets a specified defined criteria. A participant with multiple occurrences of DLTs under one treatment is counted only once in the Adverse Event category for that treatment. A participant with multiple DLTs within a primary system organ class is counted only once in the total row.
Time Frame: up to day 21 after the patient's first dose; cycle = within the first 21 days of patient's first dose
Population: The dose determining analysis set (DDS) consisted of all patients from the Safety set who either met the minimum exposure criterion and had sufficient safety evaluations or discontinued earlier due to DLT in the escalation phase.
Measure: Number; unit: Participants
Arm/Group | Fasted: Ceritinib 300 mg/m2 | Fasted: Ceritinib 450 mg/m2 | Fasted: Ceritinib 510 mg/m2 | Fasted: Ceritinib 560 mg/m2 | Fed: Ceritinib 320 mg/m2 | Fed: Ceritinib 400 mg/m2 | Fed: Ceritinib 500 mg/m2
Number analyzed (Participants) | 4 | 12 | 6 | 2 | 4 | 4 | 5
Participants
  Investigations: Alanine aminotransferase incr. | 0 | 0 | 0 | 1 | 0 | 1 | 0
  Gastrointestinal disorders: abdominal pain | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Gastrointestinal disorders: Influenza | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Total DLTs | 0 | 0 | 0 | 2 | 0 | 1 | 1
Statistical Analysis 1: Comparison: Fasted: Ceritinib 300 mg/m2 vs Fasted: Ceritinib 450 mg/m2 vs Fasted: Ceritinib 510 mg/m2 vs Fasted: Ceritinib 560 mg/m2; Test type: Other; MTD/RDE = 510
Statistical Analysis 2: Comparison: Fed: Ceritinib 320 mg/m2 vs Fed: Ceritinib 400 mg/m2 vs Fed: Ceritinib 500 mg/m2; Test type: Other; MTD/RDE = 500

2. Secondary Outcome: Summary of Best Overall Response by Overall Response Rate (ORR) Per Investigator Assessment
Description: ORR is the percentage of participants with a best overall response of complete response (CR) or partial response (PR). ORR was assessed per Investigator as per RECIST 1.1 in participants with neuroblastoma and other solid tumors, and by International Working Group (IWG) criteria in patients with lymphoma. Per RECIST 1.1 (for neuroblastoma & other solid tumors): CR: disappearance of all non-nodal target lesions. In addition, any pathological lymph nodes assigned as target lesions must have a reduction in short axis to < 10 mm. PR: at least a 30% decrease in the sum of diameter of all target lesion, taking as reference the baseline sum diameters. Per IWG criteria (for patients with lymphoma): CR: normalization of all index nodal lesions or complete disappearance of all index extranodal lesions. PR: at least 50% decrease from baseline in the sum of diameters of all index lesions.
Time Frame: 30 months
Population: Full Analysis Set (FAS)/Maximum Tolerated Dose MTD)/Recommended dose for expansion (RDE): Results are presented only for patients who received at least 1 dose of ceritinib in either of the 2 MTD/RDE groups and were based on combining data from across the dose-escalation & dose-expansion phases, & summarized according to primary diagnosis of tumor.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- ALK-activated Neuroblastoma: Participants with ALK-activated neuroblastoma enrolled in the expansion part of the study and were given ceritinib once daily, continuously
- ALK-activated Inflammatory Myofibroblastic Tumors (IMT): Participants with ALK-activated IMT enrolled in the expansion part of the study who were given ceritinib once daily, continuously
- ALK-activated Anaplastic Large Cell Lymphoma (ALCL): Participants with ALK-activated ALCL enrolled in the expansion part of the study who were given ceritinib once daily, continuously
- ALK-activated Other: Participants with other ALK-activated tumors enrolled in the expansion part of the study who were given ceritinib once daily, continuously
Arm/Group | ALK-activated Neuroblastoma | ALK-activated Inflammatory Myofibroblastic Tumors (IMT) | ALK-activated Anaplastic Large Cell Lymphoma (ALCL) | ALK-activated Other
Number analyzed (Participants) | 30 | 10 | 8 | 7
percentage of participants | 20.0 [7.7 to 38.6] | 70.0 [34.8 to 93.3] | 75.0 [34.9 to 96.8] | 14.3 [0.4 to 57.9]

3. Secondary Outcome: Duration of Response (DoR) Per Investigator Assessment
Description: DOR is defined as the time from first documented response (PR or CR) to the date of first documented disease progression (PD) or death due to any cause. DOR was assessed per Investigator as per RECIST 1.1 in participants with neuroblastoma and other solid tumors, and by International Working Group (IWG) criteria in patients with lymphoma. Per RECIST 1.1 (for neuroblastoma & other solid tumors): CR: disappearance of all non-nodal target lesions. In addition, any pathological lymph nodes assigned as target lesions must have a reduction in short axis to < 10 mm. PR: at least a 30% decrease in the sum of diameter of all target lesion, taking as reference the baseline sum diameters. Per IWG criteria (for patients with lymphoma): CR: normalization of all index nodal lesions or complete disappearance of all index extranodal lesions. PR: at least 50% decrease from baseline in the sum of diameters of all index lesions.
Time Frame: 30 months
Population: Full Analysis Set/MTD/RDE patients with confirmed CR or PR): Efficacy results are presented only for patients with confirmed CR or PR who received at least 1 dose of ceritinib in either of the 2 MTD/RDE groups & were based on combining data from across the dose-escalation & dose-expansion phases, & summarized according to primary tumor diagnosis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | ALK-activated Neuroblastoma | ALK-activated Inflammatory Myofibroblastic Tumors (IMT) | ALK-activated Anaplastic Large Cell Lymphoma (ALCL) | ALK-activated Other
Number analyzed (Participants) | 6 | 7 | 6 | 1
months | 15.0 [5.8 to 22.2] | NA [3.5 to NA] — N/A: Median not reached for subjects with ALCL, IMT & Other tumor types as most of the subjects did not have a DOR event (progression or death). | NA [2.8 to NA] — N/A: Median not reached for subjects with ALCL, IMT & Other tumor types as most of the subjects did not have a DOR event (progression or death). | NA [NA to NA] — N/A: Median not reached for subjects with ALCL, IMT & Other tumor types as most of the subjects did not have a DOR event (progression or death).

4. Secondary Outcome: Progression Free Survival (PFS) Based on Investigator Assessment
Description: PFS is the time from date of randomization/start of treatment to the date of event defined as the first documented progression or death due to any cause. PFS was assessed per Investigator as per RECIST 1.1 in participants with neuroblastoma and other solid tumors, and by International Working Group (IWG) criteria in patients with lymphoma. Per RECIST 1.1 (for neuroblastoma & other solid tumors): CR: disappearance of all non-nodal target lesions. In addition, any pathological lymph nodes assigned as target lesions must have a reduction in short axis to < 10 mm. PR: at least a 30% decrease in the sum of diameter of all target lesion, taking as reference the baseline sum diameters. Per IWG criteria (for patients with lymphoma): CR: normalization of all index nodal lesions or complete disappearance of all index extranodal lesions. PR: at least 50% decrease from baseline in the sum of diameters of all index lesions.
Time Frame: 30 months
Population: Full Analysis Set (FAS)/MTD/RDE: Efficacy results are presented only for patients who received at least 1 dose of ceritinib in either of the two MTD/RDE groups and were based on combining data from across the dose-escalation & dose-expansion phases, & summarized according to primary diagnosis of tumor.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | ALK-activated Neuroblastoma | ALK-activated Inflammatory Myofibroblastic Tumors (IMT) | ALK-activated Anaplastic Large Cell Lymphoma (ALCL) | ALK-activated Other
Number analyzed (Participants) | 30 | 10 | 8 | 7
months | 2.4 [1.2 to 6.8] | NA [1.2 to NA] — N/A: The median was not reached for subjects with IMT and ALCL | NA [4.1 to NA] — N/A: The median was not reached for subjects with IMT and ALCL | 1.9 [1.2 to NA] — N/A: The median was not reached for subjects with IMT and ALCL

5. Secondary Outcome: Plasma Concentration Time Profiles by Treatment Group in Escalation Phase
Description: Characterize single and multiple-dose PK of LDK378 in pediatric patients. Only PK plasma concentrations with non-missing sampling date and time, and for which the last dose date and time prior to the PK sample draw are non-missing, were included in the PK analysis.
Time Frame: 0hr pre-dose, 2hrs post-dose, 4hrs post-dose, 6hrs post-dose & 24hrs post-dose in Cycle1 Day1 & Cycle 2 day 1; 0hr pre-dose in Cycle 1 Day 15, Cycle 2 Day1, Cycle 2 Day 2, Cycle 3 day 1 & Cycle 4 Day 1
Population: The PK analysis set (PAS) consisted of all patients who received at least one dose of ceritinib and had at least one evaluable PK sample.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Fasted: Ceritinib 300 mg/m2 | Fasted: Ceritinib 450 mg/m2 | Fasted: Ceritinib 510 mg/m2 | Fasted: Ceritinib 560 mg/m2 | Fed: Ceritinib 320 mg/m2 | Fed: Ceritinib 400 mg/m2 | Fed: Ceritinib 500 mg/m2
Number analyzed (Participants) | 5 | 12 | 6 | 2 | 4 | 5 | 5
ng/mL
  Cycle1 Day1 (C1D1) 0 hr pre-dose | 0.0 (0.0) | 0.0 (0.0) | 0.0 (0.0) | 0.0 (0.0) | 0.0 (0.0) | 0.0 (0.0) | 0.0 (0.0)
  C1D1 2 hrs post-dose: number analyzed (Participants) | 5 | 11 | 6 | 2 | 4 | 5 | 5
  C1D1 2 hrs post-dose | 104 (97.9) | 99.0 (94.7) | 112 (90.6) | 126 (0.6) | 52.4 (138.1) | 197 (58.3) | 72.5 (82.3)
  C1D1 4 hrs post-dose: number analyzed (Participants) | 5 | 11 | 6 | 2 | 4 | 5 | 5
  C1D1 4 hrs post-dose | 216 (39.6) | 233 (69.0) | 250 (93.5) | 350 (54.7) | 166 (92.8) | 311 (28.1) | 153 (34.1)
  C1D1 6 hrs post-dose: number analyzed (Participants) | 5 | 11 | 6 | 2 | 4 | 5 | 4
  C1D1 6 hrs post-dose | 227 (33.8) | 245 (78.1) | 245 (97.2) | 423 (74.2) | 275 (35.3) | 318 (36.7) | 168 (68.9)
  C1D1 24 hrs post-dose: number analyzed (Participants) | 5 | 11 | 6 | 2 | 4 | 5 | 4
  C1D1 24 hrs post-dose | 130 (66.3) | 141 (89.9) | 86.4 (117.2) | 268 (73.6) | 98.5 (63.7) | 126 (107.7) | 161 (111.3)
  C1D2 0 hr pre-dose: number analyzed (Participants) | 5 | 11 | 6 | 2 | 4 | 5 | 4
  C1D2 0 hr pre-dose | 130 (66.3) | 141 (89.9) | 86.4 (117.2) | 268 (73.6) | 98.5 (63.7) | 126 (107.7) | 161 (111.3)
  C1D15 0 hr pre-dose: number analyzed (Participants) | 5 | 12 | 6 | 2 | 3 | 4 | 5
  C1D15 0 hr pre-dose | 193 (99.6) | 618 (64.6) | 537 (49.9) | 942 (5.1) | 262 (118.4) | 379 (119.2) | 461 (76.3)
  C2D1 0 hr pre-dose: number analyzed (Participants) | 5 | 12 | 5 | 2 | 3 | 4 | 3
  C2D1 0 hr pre-dose | 169 (299.5) | 661 (53.5) | 672 (45.4) | 695 (152.7) | 218 (103.7) | 429 (73.8) | 655 (12.4)
  C2D1 2 hrs post-dose: number analyzed (Participants) | 5 | 12 | 5 | 2 | 3 | 4 | 3
  C2D1 2 hrs post-dose | 287 (85.4) | 687 (61.6) | 801 (45.9) | 662 (99.6) | 196 (112.4) | 475 (96.6) | 718 (21.1)
  C2D1 4 hrs post-dose: number analyzed (Participants) | 5 | 12 | 5 | 2 | 3 | 4 | 3
  C2D1 4 hrs post-dose | 386 (47.6) | 810 (51.9) | 1000 (30.4) | 1230 (30.1) | 262 (133.9) | 631 (86.6) | 744 (13.2)
  C2D1 6 hrs post-dose: number analyzed (Participants) | 5 | 12 | 5 | 2 | 3 | 4 | 2
  C2D1 6 hrs post-dose | 426 (38.4) | 852 (47.8) | 898 (37.6) | 1260 (16.4) | 300 (130.3) | 648 (105.5) | 786 (7.7)
  C2D1 24 hrs post-dose: number analyzed (Participants) | 5 | 12 | 5 | 2 | 3 | 4 | 5
  C2D1 24 hrs post-dose | 247 (46.9) | 651 (53.7) | 714 (40.8) | 847 (72.2) | 194 (106.5) | 411 (147.3) | 448 (43.9)
  C2D2 0 hr pre-dose: number analyzed (Participants) | 5 | 12 | 5 | 2 | 3 | 4 | 5
  C2D2 0 hr pre-dose | 247 (46.9) | 651 (53.7) | 714 (40.8) | 847 (72.2) | 194 (106.5) | 411 (147.3) | 448 (43.9)
  C3D1 0 hr pre-dose: number analyzed (Participants) | 2 | 8 | 4 | 1 | 2 | 1 | 5
  C3D1 0 hr pre-dose | 399 (94.4) | 810 (34.3) | 415 (117.7) | 1320 (0.0) | 167 (218.3) | 328 (0.0) | 433 (128.5)
  C4D1 0 hr pre-dose: number analyzed (Participants) | 2 | 8 | 4 | 1 | 1 | 1 | 3
  C4D1 0 hr pre-dose | 503 (35.1) | 960 (36.2) | 321 (874.8) | 857 (0.0) | 403 (0.0) | 1320 (0.0) | 658 (27.0)

6. Secondary Outcome: Plasma Concentration Time Profiles by Treatment Group in Expansion Phase
Description: as for outcome 5
Time Frame: 0hr pre-dose Cycle 1 Day 1, cycle 1 Day 15; 0hr pre-dose, 2hrs post-dose, 4hrs post-dose, 6hrs post-dose & 24hrs post-dose in Cycle2 Day1; 0hr pre-dose in Cycle2 Day2, Cycle 3 Day 1 & Cycle 4 Day 1
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Fasted: Ceritinib 300 mg/m2 | Fasted: Ceritinib 450 mg/m2 | Fasted: Ceritinib 510 mg/m2 | Fasted: Ceritinib 560 mg/m2 | Fed: Ceritinib 320 mg/m2 | Fed: Ceritinib 400 mg/m2 | Fed: Ceritinib 500 mg/m2
Number analyzed (Participants) | 0 | 0 | 7 | 0 | 0 | 0 | 16
ng/mL
  C1D1 0 hr pre-dose: number analyzed (Participants) | 0 | 0 | 6 | 0 | 0 | 0 | 9
  C1D1 0 hr pre-dose |  |  | 0.0 (0.0) |  |  |  | 0.0 (0.0)
  C1D15 0 hr post-dose: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0 | 0
  C1D15 0 hr post-dose |  |  | 1190 (0.0) |  |  |  |
  C2D1 0 hr pre-dose |  |  | 529 (365.4) |  |  |  | 627 (93.6)
  C2D1 2 hrs post-dose: number analyzed (Participants) | 0 | 0 | 7 | 0 | 0 | 0 | 15
  C2D1 2 hrs post-dose |  |  | 798 (69.0) |  |  |  | 729 (72.3)
  C2D1 4 hrs post-dose: number analyzed (Participants) | 0 | 0 | 7 | 0 | 0 | 0 | 14
  C2D1 4 hrs post-dose |  |  | 863 (65.2) |  |  |  | 828 (47.9)
  C2D1 6 hrs post-dose: number analyzed (Participants) | 0 | 0 | 7 | 0 | 0 | 0 | 15
  C2D1 6 hrs post-dose |  |  | 939 (71.4) |  |  |  | 870 (52.6)
  C2D1 24 hrs post-dose: number analyzed (Participants) | 0 | 0 | 6 | 0 | 0 | 0 | 14
  C2D1 24 hrs post-dose |  |  | 615 (119.9) |  |  |  | 596 (75.5)
  C2D2 0 hr pre-dose: number analyzed (Participants) | 0 | 0 | 6 | 0 | 0 | 0 | 14
  C2D2 0 hr pre-dose |  |  | 615 (119.9) |  |  |  | 596 (75.5)
  C3D1 0 hr pre-dose: number analyzed (Participants) | 0 | 0 | 5 | 0 | 0 | 0 | 14
  C3D1 0 hr pre-dose |  |  | 836 (60.4) |  |  |  | 573 (134.2)
  C4D1 0 hr pre-dose: number analyzed (Participants) | 0 | 0 | 5 | 0 | 0 | 0 | 12
  C4D1 0 hr pre-dose |  |  | 834 (78.8) |  |  |  | 622 (96.5)

7. Secondary Outcome: Pharmacokinetics (PK) Parameters: AUC0 - 24h & AUClast in Cycle 1 Day 1 - Dose Escalation Phase (Single Dose)
Description: Characterize single and multiple-dose PK of LDK378 in pediatric patients. AUC: Area under the plasma (serum, or blood) concentration versus time curve AUClast: Area under the concentration-time curve from time zero to the last measureable concentration time AUC0-24h: Area under the plasma concentration-time curve t=0-24 h
Time Frame: 0hr pre-dose, 2, 4, 6 & 24hrs post-dose
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*ng/mL
Arm/Group | Fasted: Ceritinib 300 mg/m2 | Fasted: Ceritinib 450 mg/m2 | Fasted: Ceritinib 510 mg/m2 | Fasted: Ceritinib 560 mg/m2 | Fed: Ceritinib 320 mg/m2 | Fed: Ceritinib 400 mg/m2 | Fed: Ceritinib 500 mg/m2
Number analyzed (Participants) | 5 | 10 | 3 | 1 | 3 | 4 | 3
hr*ng/mL
  AUC0-24h: number analyzed (Participants) | 4 | 3 | 2 | 0 | 1 | 1 | 2
  AUC0-24h | 3920 (39.9) | 5220 (58.0) | 8750 (11.1) |  | 5720 (0.0) | 7272 (0.0) | 4730 (59.4)
  AUClast: number analyzed (Participants) | 5 | 9 | 3 | 1 | 3 | 4 | 3
  AUClast | 4260 (39.3) | 4350 (91.8) | 7670 (24.5) | 4860 (0.0) | 3730 (48.6) | 5760 (49.1) | 4940 (32.6)

8. Secondary Outcome: Pharmacokinetics (PK) Parameters: AUC0 - 24h & AUClast in Cycle 2 Day 1 - Dose Escalation Phase (Single Dose)
Description: Characterize single and multiple-dose PK of LDK378 in pediatric patients. AUC: Area under the plasma (serum, or blood) concentration versus time curve AUClast: Area under the concentration-time curve from time zero to the last measureable concentration time; AUC0-24h: Area under the plasma concentration-time curve t=0-24 h
Time Frame: 0hr pre-dose, 2, 4, 6 & 24hrs post-dose
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*ng/mL
Arm/Group | Fasted: Ceritinib 300 mg/m2 | Fasted: Ceritinib 450 mg/m2 | Fasted: Ceritinib 510 mg/m2 | Fasted: Ceritinib 560 mg/m2 | Fed: Ceritinib 320 mg/m2 | Fed: Ceritinib 400 mg/m2 | Fed: Ceritinib 500 mg/m2
Number analyzed (Participants) | 5 | 12 | 5 | 2 | 3 | 4 | 2
hr*ng/mL
  AUC0-24h: number analyzed (Participants) | 5 | 7 | 2 | 2 | 1 | 1 | 1
  AUC0-24h | 8160 (44.0) | 16900 (59.1) | 21000 (20.8) | 25300 (39.2) | 2100 (0.0) | 30500 (0.0) | 16500 (0.0)
  AUClast | 8210 (44.3) | 18000 (50.0) | 17200 (51.2) | 25600 (39.0) | 5840 (118.4) | 125000 (113.2) | 16700 (1.8)

9. Secondary Outcome: Pharmacokinetics (PK) Parameters: AUC0 - 24h & AUClast in Cycle 2 Day 1 - Dose Expansion Phase (Multiple Dose)
Description: Characterize single and multiple-dose PK of LDK378 in pediatric patients. In this phase ceritinib was expanded at 500mg/m2 fed and 510mg/m2 fasted administered orally once daily and was assessed only at steady state, Cycle 2 Day 1.
  AUC: Area under the plasma (serum, or blood) concentration versus time curve AUClast: Area under the plasma (serum, or blood) concentration versus time curverea under the concentration-time curve from time zero to the last measureable concentration time AUC0-24h: Area under the plasma concentration-time curve t=0-24 h
Time Frame: 0hr pre-dose, 2, 4, 6 & 24hrs post-dose
Population: The PK analysis set (PAS), MTD/RDE consisted of all patients who received at least one dose of ceritinib and had at least one evaluable PK sample.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*ng/mL
Arm/Group | Fasted: Ceritinib 510 mg/m2 | Fed: Ceritinib 500 mg/m2
Number analyzed (Participants) | 4 | 14
hr*ng/mL
  AUC0-24h: number analyzed (Participants) | 0 | 6
  AUC0-24h |  | 15900 (93.8)
  AUClast | 24100 (38.9) | 16100 (61.2)

10. Secondary Outcome: PK Parameter: Cmax in Cycle 1 Day 1 - Dose Escalation Phase (Single Dose)
Description: Characterize single and multiple-dose PK of LDK378 in pediatric patients. Cmax: Maximum (peak) concentration of drug
Time Frame: 0hr pre-dose, 2, 4, 6 & 24hrs post-dose
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Fasted: Ceritinib 300 mg/m2 | Fasted: Ceritinib 450 mg/m2 | Fasted: Ceritinib 510 mg/m2 | Fasted: Ceritinib 560 mg/m2 | Fed: Ceritinib 320 mg/m2 | Fed: Ceritinib 400 mg/m2 | Fed: Ceritinib 500 mg/m2
Number analyzed (Participants) | 5 | 10 | 3 | 1 | 3 | 4 | 3
ng/mL | 258 (39.0) | 270 (82.1) | 537 (22.2) | 265 (0.0) | 251 (37.0) | 341 (34.2) | 204 (54.6)

11. Secondary Outcome: PK Parameter: Cmax in Cycle 2 Day 1 - Dose Escalation Phase (Single Dose)
Description: Characterize single and multiple-dose PK of LDK378 in pediatric patients. Cmax: Maximum (peak) concentration of drug.
Time Frame: 0hr pre-dose, 2, 4, 6 & 24hrs post-dose
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Fasted: Ceritinib 300 mg/m2 | Fasted: Ceritinib 450 mg/m2 | Fasted: Ceritinib 510 mg/m2 | Fasted: Ceritinib 560 mg/m2 | Fed: Ceritinib 320 mg/m2 | Fed: Ceritinib 400 mg/m2 | Fed: Ceritinib 500 mg/m2
Number analyzed (Participants) | 5 | 12 | 5 | 2 | 3 | 4 | 2
ng/mL | 427 (38.5) | 870 (48.7) | 1020 (32.1) | 1300 (21.4) | 300 (130.3) | 674 (93.8) | 804 (10.4)

12. Secondary Outcome: PK Parameter: Cmax in Cycle 2 Day 1 - Dose Expansion Phase (Multiple Dose)
Description: Characterize single and multiple-dose PK of LDK378 in pediatric patients. In this phase ceritinib was expanded at 500mg/m2 fed and 510mg/m2 fasted administered orally once daily and was assessed only at steady state, Cycle 2 Day 1.
  Cmax: Maximum (peak) concentration of drug
Time Frame: 0hr pre-dose, 2, 4, 6 & 24hrs post-dose
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Fasted: Ceritinib 510 mg/m2 | Fed: Ceritinib 500 mg/m2
Number analyzed (Participants) | 4 | 14
ng/mL | 1220 (40.2) | 890 (50.9)

13. Secondary Outcome: PK Parameter: Tmax in Cycle 1 Day 1 - Dose Escalation Phase (Single Dose)
Description: Characterize single and multiple-dose PK of LDK378 in pediatric patients. Tmax: The time to reach maximum plasma concentration
Time Frame: 0hr pre-dose, 2, 4, 6 & 24hrs post-dose
Population: as for outcome 5
Measure: Median (Full Range); unit: hour (hr)
Arm/Group | Fasted: Ceritinib 300 mg/m2 | Fasted: Ceritinib 450 mg/m2 | Fasted: Ceritinib 510 mg/m2 | Fasted: Ceritinib 560 mg/m2 | Fed: Ceritinib 320 mg/m2 | Fed: Ceritinib 400 mg/m2 | Fed: Ceritinib 500 mg/m2
Number analyzed (Participants) | 5 | 10 | 3 | 1 | 3 | 4 | 3
hour (hr) | 4.20 [1.90 to 24.0] | 4.25 [0.00 to 6.10] | 4.30 [4.10 to 6.00] | 6.10 [6.10 to 6.10] | 6.10 [5.70 to 6.30] | 6.00 [4.30 to 6.20] | 5.80 [4.10 to 6.10]

14. Secondary Outcome: PK Parameter: Tmax in Cycle 2 Day 1 - Dose Escalation Phase (Single Dose)
Description: as for outcome 13
Time Frame: 0hr pre-dose, 2, 4, 6 & 24hrs post-dose
Population: as for outcome 5
Measure: Median (Full Range); unit: hour (hr)
Arm/Group | Fasted: Ceritinib 300 mg/m2 | Fasted: Ceritinib 450 mg/m2 | Fasted: Ceritinib 510 mg/m2 | Fasted: Ceritinib 560 mg/m2 | Fed: Ceritinib 320 mg/m2 | Fed: Ceritinib 400 mg/m2 | Fed: Ceritinib 500 mg/m2
Number analyzed (Participants) | 5 | 12 | 5 | 2 | 3 | 4 | 2
hour (hr) | 6.00 [4.10 to 6.70] | 5.10 [2.00 to 6.60] | 4.00 [2.10 to 6.00] | 3.95 [0.00 to 6.70] | 5.90 [5.80 to 6.10] | 6.00 [4.00 to 6.10] | 2.20 [2.00 to 2.40]

15. Secondary Outcome: PK Parameter: Tmax in Cycle 2 Day 1 - Dose Expansion Phase (Multiple Dose)
Description: Characterize single and multiple-dose PK of LDK378 in pediatric patients. In this phase ceritinib was expanded at 500mg/m2 fed and 510mg/m2 fasted administered orally once daily and was assessed only at steady state, Cycle 2 Day 1.
  Characterize single and multiple-dose PK of LDK378 in pediatric patients. Tmax: The time to reach maximum plasma concentration
Time Frame: 0hr pre-dose, 2, 4, 6 & 24hrs post-dose
Population: as for outcome 9
Measure: Median (Full Range); unit: hour (hr)
Arm/Group | Fasted: Ceritinib 510 mg/m2 | Fed: Ceritinib 500 mg/m2
Number analyzed (Participants) | 4 | 14
hour (hr) | 6.20 [3.80 to 23.8] | 5.90 [1.90 to 23.6]

16. Secondary Outcome: PK Parameter: Racc in Dose Escalation Phase Cycle 2 Day 1
Description: Characterize single and multiple-dose PK of LDK378 in pediatric patients. Racc: Accumulation ratio
Time Frame: 0hr pre-dose, 2, 4, 6 & 24hrs post-dose
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Fasted: Ceritinib 300 mg/m2 | Fasted: Ceritinib 450 mg/m2 | Fasted: Ceritinib 510 mg/m2 | Fasted: Ceritinib 560 mg/m2 | Fed: Ceritinib 320 mg/m2 | Fed: Ceritinib 400 mg/m2 | Fed: Ceritinib 500 mg/m2
Number analyzed (Participants) | 5 | 12 | 5 | 2 | 3 | 4 | 2
ratio | 1.93 (64.2) | 5.50 (30.3) | 2.56 (0.0) | 6.86 (0.0) | 0.533 (0.0) | 3.41 (0.0) | 3.62 (0.0)

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected from first dose of study treatment until end of study treatment plus 30 days post treatment, up to maximum duration of 63.7 months.
Description: AE is any sign or symptom that occurs during the study treatment plus the 30 days post treatment
Groups:
- Fasted Ceritinib 300mg/m2: Participants in the fasted group who took 300 mg of ceritinib
- Fasted Ceritinib 450mg/m2: Participants in the fasted group who took 450 mg of ceritinib
- Fasted Ceritinib 510mg/m2: Participants in the fasted group who took 510 mg of ceritinib
- Fasted Ceritinib 560mg/m2: Participants in the fasted group who took 560 mg of ceritinib
- Fed Ceritinib 320mg/m2: Participants in the fed group who took 320 mg of ceritinib
- Fed Ceritinib 400mg/m2: Participants in the fed group who took 400 mg of ceritinib
- Fed Ceritinib 500mg/m2: Participants in the fed group who took 500 mg of ceritinib
- Fasted+Fed All Patients: All participants in the Fasted and Fed groups
Arm/Group | Fasted Ceritinib 300mg/m2 | Fasted Ceritinib 450mg/m2 | Fasted Ceritinib 510mg/m2 | Fasted Ceritinib 560mg/m2 | Fed Ceritinib 320mg/m2 | Fed Ceritinib 400mg/m2 | Fed Ceritinib 500mg/m2 | Fasted+Fed All Patients
All-Cause Mortality (participants affected / at risk) | 1/5 | 1/12 | 2/13 | 0/2 | 2/4 | 1/5 | 5/42 | 12/83
Serious Adverse Events (participants affected / at risk) | 1/5 | 4/12 | 8/13 | 2/2 | 3/4 | 1/5 | 21/42 | 40/83
Other Adverse Events (participants affected / at risk) | 5/5 | 12/12 | 13/13 | 2/2 | 4/4 | 5/5 | 42/42 | 83/83
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fasted Ceritinib 300mg/m2 (N=5) | Fasted Ceritinib 450mg/m2 (N=12) | Fasted Ceritinib 510mg/m2 (N=13) | Fasted Ceritinib 560mg/m2 (N=2) | Fed Ceritinib 320mg/m2 (N=4) | Fed Ceritinib 400mg/m2 (N=5) | Fed Ceritinib 500mg/m2 (N=42) | Fasted+Fed All Patients (N=83)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2
Febrile bone marrow aplasia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Cardiac failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Pericarditis (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 1 | 1 | 1 | 0 | 1 | 5
Ascites (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Dental caries (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Small intestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Subileus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Chest pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 2
General physical health deterioration (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Multiple organ dysfunction syndrome (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 3 | 6
Acute hepatic failure (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Hepatotoxicity (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Device related infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 4
Ear infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Encephalitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Enterovirus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2
Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3
Metapneumovirus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Pneumonia viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Pyelonephritis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3
Septic shock (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Staphylococcal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Tonsillitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Wound infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1 | 1 | 0 | 0 | 0 | 2 | 4
Amylase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 2 | 0 | 0 | 0 | 1 | 4
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
C-reactive protein increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Lipase increased (Investigations) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 2
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Hemiplegia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Seizure (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2
Suicide attempt (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 2
Bronchopleural fistula (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Hypotension (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Fasted Ceritinib 300mg/m2 (N=5) | Fasted Ceritinib 450mg/m2 (N=12) | Fasted Ceritinib 510mg/m2 (N=13) | Fasted Ceritinib 560mg/m2 (N=2) | Fed Ceritinib 320mg/m2 (N=4) | Fed Ceritinib 400mg/m2 (N=5) | Fed Ceritinib 500mg/m2 (N=42) | Fasted+Fed All Patients (N=83)
Anaemia (Blood and lymphatic system disorders) | 1 | 3 | 3 | 1 | 3 | 0 | 11 | 22
Bone marrow disorder (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 2
Leukopenia (Blood and lymphatic system disorders) | 1 | 0 | 2 | 0 | 0 | 0 | 5 | 8
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 1 | 1 | 3 | 0 | 0 | 0 | 5 | 10
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 2 | 2 | 2 | 2 | 0 | 11 | 19
Left ventricular dysfunction (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Palpitations (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 2
Pericardial effusion (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 2
Tachycardia (Cardiac disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 2 | 4
Ear pain (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 3 | 4
External ear inflammation (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Hypoacusis (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Delayed puberty (Endocrine disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Hypothyroidism (Endocrine disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 2
Eye pain (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Eye swelling (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Ocular discomfort (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vision blurred (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 3 | 6 | 6 | 2 | 2 | 1 | 22 | 42
Abdominal pain upper (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 1 | 1 | 3 | 7
Anal fissure (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Anal incontinence (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Anal inflammation (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 3 | 2 | 2 | 1 | 1 | 1 | 4 | 14
Diarrhoea (Gastrointestinal disorders) | 4 | 12 | 10 | 2 | 2 | 3 | 32 | 65
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 4 | 6
Flatulence (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 1 | 1 | 4
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Gingival pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Haematemesis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Haematochezia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 2 | 8 | 10 | 1 | 2 | 3 | 21 | 47
Odynophagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3
Proctalgia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Stomatitis (Gastrointestinal disorders) | 1 | 1 | 0 | 1 | 0 | 0 | 3 | 6
Vomiting (Gastrointestinal disorders) | 4 | 10 | 13 | 2 | 4 | 3 | 36 | 72
Asthenia (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 9 | 10
Catheter site pain (General disorders) | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 3
Chest pain (General disorders) | 0 | 2 | 1 | 0 | 1 | 1 | 6 | 11
Fatigue (General disorders) | 3 | 4 | 3 | 2 | 1 | 0 | 9 | 22
Gait disturbance (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
General physical health deterioration (General disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 2
Influenza like illness (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Malaise (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Oedema peripheral (General disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 4
Pyrexia (General disorders) | 3 | 4 | 6 | 1 | 0 | 1 | 20 | 35
Secretion discharge (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3
Ulcer (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Hepatomegaly (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 2
Bacterial vulvovaginitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 3
Conjunctivitis (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 0 | 3 | 5
Device related infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3
Ear infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 3
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 4
Genital candidiasis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Human herpesvirus 6 infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Influenza (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 | 2 | 4
Molluscum contagiosum (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Mycoplasma infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 2 | 1 | 2 | 0 | 1 | 0 | 4 | 10
Oral herpes (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 2
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3
Rhinitis (Infections and infestations) | 0 | 2 | 1 | 0 | 0 | 0 | 8 | 11
Sinusitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 2 | 3 | 1 | 0 | 0 | 8 | 15
Urinary tract infection (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 3
Varicella (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 2
Viral infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2
Wound infection (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 2
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 2
Hand fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Muscle injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 8 | 8 | 2 | 3 | 2 | 30 | 54
Amylase increased (Investigations) | 0 | 1 | 1 | 0 | 0 | 1 | 3 | 6
Aspartate aminotransferase increased (Investigations) | 1 | 6 | 7 | 2 | 3 | 1 | 28 | 48
Blood albumin decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 1 | 4 | 0 | 0 | 1 | 0 | 4 | 10
Blood bicarbonate decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 2
Blood bilirubin increased (Investigations) | 0 | 2 | 0 | 0 | 1 | 0 | 5 | 8
Blood creatine increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3
Blood creatine phosphokinase MB increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Blood creatinine increased (Investigations) | 2 | 4 | 1 | 0 | 0 | 0 | 11 | 18
Blood glucose increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Blood lactate dehydrogenase increased (Investigations) | 0 | 2 | 3 | 0 | 0 | 1 | 5 | 11
Blood magnesium increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3
Blood pressure increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Blood urea increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3
Blood uric acid increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 3 | 4
C-reactive protein increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 1 | 4 | 6
Electrocardiogram QT prolonged (Investigations) | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 3
Gamma-glutamyltransferase increased (Investigations) | 0 | 3 | 3 | 1 | 2 | 3 | 14 | 26
Haemoglobin decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 3
Lipase increased (Investigations) | 0 | 0 | 2 | 0 | 0 | 1 | 6 | 9
Lymphocyte count decreased (Investigations) | 0 | 1 | 1 | 0 | 0 | 0 | 2 | 4
Neutrophil count decreased (Investigations) | 0 | 1 | 1 | 0 | 1 | 0 | 2 | 5
Platelet count decreased (Investigations) | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 3
Prothrombin time prolonged (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Prothrombin time shortened (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Troponin increased (Investigations) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 2
Tumour marker increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Weight decreased (Investigations) | 1 | 2 | 3 | 1 | 0 | 0 | 6 | 13
White blood cell count decreased (Investigations) | 1 | 1 | 0 | 1 | 0 | 0 | 1 | 4
White blood cell count increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 3 | 4 | 0 | 2 | 1 | 0 | 16 | 26
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Fluid retention (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 2
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 4 | 5
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 1 | 4
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 1 | 0 | 0 | 0 | 1 | 7 | 12
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 3 | 5
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 1 | 1 | 0 | 0 | 0 | 3 | 7
Hypophosphataemia (Metabolism and nutrition disorders) | 2 | 2 | 1 | 0 | 1 | 0 | 2 | 8
Obesity (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 4 | 6
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 0 | 1 | 0 | 2 | 6
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 3
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 3
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1 | 0 | 0 | 0 | 2 | 5
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 5 | 0 | 0 | 1 | 1 | 5 | 13
Torticollis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 2 | 1 | 0 | 0 | 0 | 2 | 5
Dysaesthesia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Dysgeusia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 3 | 4 | 1 | 0 | 2 | 1 | 8 | 19
Hypertonia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Lethargy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Migraine (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Neuralgia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Somnolence (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Tremor (Nervous system disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 3
Anxiety (Psychiatric disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 3
Irritability (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Mental disorder (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Restlessness (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Sleep disorder (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Dysuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Micturition urgency (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Pollakiuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Dysmenorrhoea (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2 | 1 | 0 | 0 | 8 | 13
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 4 | 6
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 2 | 4
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 3 | 5
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 3
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 2
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 3 | 4
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Acne (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 2 | 4
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 3
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 4
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 2 | 2 | 1 | 0 | 1 | 1 | 7
Rash (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 6 | 8
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 3 | 1 | 0 | 0 | 0 | 1 | 5
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 2
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Skin irritation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Swelling face (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 2
Embolism (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Haematoma (Vascular disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 2
Hypertension (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 2
Hypotension (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Pallor (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of pooled data (i.e.,data from all sites) in clinical trial or disclosure of trial results in their entirety.

DOCUMENTS (2):
  • Study Protocol (2018-05-18): https://cdn.clinicaltrials.gov/large-docs/86/NCT01742286/Prot_000.pdf
  • Statistical Analysis Plan (2019-05-30): https://cdn.clinicaltrials.gov/large-docs/86/NCT01742286/SAP_001.pdf